CLINICAL TRIAL: NCT03302117
Title: Pulmonary and Systemic Effects of Exposure to Wood Smoke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Other Study IDs: WSIII
Record Dates: First submitted 2017-09-21; First posted 2017-10-04 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-09

CONDITIONS: Pulmonary Inflammation; Cytotoxicity
Keywords: Wood smoke; Bronchoscopy
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bronchoalevolar lavage. Endobronchial biopsies. Peripheral blood sampling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Wood smoke exposure — Healthy volunteers will exposed to filtered air alternate with wood smoke generated from incomplete wood smoke combustion to assess the local and systemic effect of theses exposures

SUMMARY:
This is study is to assess pulmonary and systemic effects of exposure to wood smoke. Healthy volunteers will be expose under two different occasion to wood smoke and filtered air under two separated occasions with an interval of 3 weeks in-between. The aim of this study was to determine whether exposure to wood smoke from incomplete combustion would elicit airway inflammation in humans.

DETAILED DESCRIPTION:
Brief Summary This is study is to assess pulmonary and systemic effects of exposure to wood smoke. Healthy volunteers will be expose under two different occasion to wood smoke and to filtered air for two hours under two separated occasions with an interval of 3 weeks in-between. The aim of this study was to determine whether exposure to wood smoke from incomplete combustion would elicit airway inflammation in humans.

Detailed description Air pollution is associate with increased pulmonary and cardiovascular mobility and mortality. UNICEF recently published a report highlighting the health effects of air pollution from a global perspective, with particular focus on pediatrics population. Overall, air pollution is estimated to cause about 7 million deaths each year in the world, of which about 600,000 of these apply to children under 5 years (1). Indoor and outdoor air pollutants are the 3rd and 9th most common cause of death. Nearly 3 billion people are dependent on biomass for daily needs, Exposure to wood smoke has been linked to elevated asthma prevalence, increased asthma symptoms in children and adults, as well as higher hospital admissions due to asthma attacks. The association between long-term indoor wood smoke exposure and the development and worsening of chronic obstructive pulmonary disease has been shown to be strong in many epidemiological studies (2,3), and the risk for chronic obstructive pulmonary disease development has been estimated to be more than doubled for solid fuel smoke compared with smoke from other types of fuels (4). Exposure to smoke from combustion of wood and other biomass fuels has also been shown to increase the risk for acute and chronic lower respiratory tract infections, including pneumonias and tuberculosis. The aim of the current study was to further characterize the respiratory and systemic effects of exposure to wood smoke emitted from incomplete soot-rich combustion in a wood stove.

The study will be performed in a randomized, double blind, crossover fashion. Twenty healthy subjects will be exposed on two occasions, under well-controlled situations, to filtered air and wood smoke in an exposure chamber at Thermochemical Energy Conversion Laboratory at Umeå University. The chamber is made of stainless steel, has a volume of a 15.3 m3 and an air exchange rate of around three times per hour and has been previously described (5). The mean particle mass concentration of wood smoke will be 450 μg/m3. The exposures will last for two hours, during which the subject will perform intermittent exercise on a bicycle ergometer, alternate with rest at 15-minute intervals, to achieve an average minute ventilation of 20 L/min/m2 body surface. During the exposures, symptoms well be recorded according to the modified Borg scale, as described previously (6). Spirometry and impulse oscillometry system (IOS) will be used to assess the lung function at baseline and immediately after each exposure. Bronchoscopy will be performed 6 hours after each exposure. Differential cell counts and soluble components will be analyzed in peripheral blood sampling at baseline and 6 hours after each exposure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Non-smoker
* Non-allergic

Exclusion Criteria:

* Diabetes Mellitus
* Renal failure
* Ischemic heart disease
* History of hematological disease
* Previous smoking.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Twenty healthy volunteers (age 20-40, all never smokers) will included. All subjects undergo a physical examination, baseline blood count and renal function assessment, spirometry (FEV1, VC and FEV1/VC) and 12 lead electrocardiogram prior to inclusion. All must be free of airway infection for at least 6 weeks prior to participation. The study was approved by the regional ethical review board and performed in accordance with the declaration of Helsinki. All subjects should give their written informed consent.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-06-14 (Actual); Primary Completion 2018-02-08 (Estimated); Study Completion 2018-02-08 (Estimated)

PRIMARY OUTCOMES:
Pulmonary inflammation | Bronchoscopy will be done 6 hours after each exposure.
  Flexible bronchoscopy will done to obtain bronchoalveolar lavage to assess the inflammatory responses by measurement of cell differential counts and cytokines level.
Pulmonary cytotoxicity | Bronchoscopy will be done 6 hours after each exposure.
  Bronchoalveolar lavage will be examined for signs of cytotoxicity by measurement of cell death and apoptosis markers.
Inflammatory changes in endobronchial biopsies | Bronchoscopy will be done 6 hours after each exposure and the processing of the immunohistochemistry method will start immediately after each bronchoscopy
  Endobronchial biopsies will be obtained by using flexible bronchoscopy. The biopsies will be stained by using immunohistochemistry method for assessing the inflammatory responses after each exposures

SECONDARY OUTCOMES:
Systemic inflammatory responses | Before and 6 hour after each exposure
  Peripheral blood samples will be centrifuged at 3,000xg for 30 min at 4 Celsius and then plasma will be removed and frozen at -80 Celsius for further analysis. Plasma samples will be analysed for markers of acute inflammation: Interleukin 6 (IL-6), tumor necrosis factor-alpha (TNF-α), soluble Intercellular Adhesion Molecule-1 (sICAM-1) and club cell secretory protein 16 (CC16, formerly called clara cell protein 16) using ELISA kits.
Lung function test | At baseline, immediately after and 6 hours after each exposure
  Assessment of lung function by using using a spirometer (Jaeger spirometer, Germany). The tests were performed according to the guidelines of the American Thoracic Society. An new method will used here also by using impulse oscillometry system (IOS).

CONTACTS AND LOCATIONS:
Overall Officials: Ala Muala, MD, PhD, Principal Investigator — Department for Public Health and Clinical Medicine
Locations (1):
- Department for Public Health and Clinical Medicine, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friedrich MJ. UNICEF Reports on the Impact of Air Pollution on Children. JAMA. 2017 Jan 17;317(3):246. doi: 10.1001/jama.2016.19034. No abstract available. PMID 28114563
- [Background] Po JY, FitzGerald JM, Carlsten C. Respiratory disease associated with solid biomass fuel exposure in rural women and children: systematic review and meta-analysis. Thorax. 2011 Mar;66(3):232-9. doi: 10.1136/thx.2010.147884. Epub 2011 Jan 19. PMID 21248322
- [Background] Hu G, Zhou Y, Tian J, Yao W, Li J, Li B, Ran P. Risk of COPD from exposure to biomass smoke: a metaanalysis. Chest. 2010 Jul;138(1):20-31. doi: 10.1378/chest.08-2114. Epub 2010 Feb 5. PMID 20139228
- [Background] Kurmi OP, Semple S, Simkhada P, Smith WC, Ayres JG. COPD and chronic bronchitis risk of indoor air pollution from solid fuel: a systematic review and meta-analysis. Thorax. 2010 Mar;65(3):221-8. doi: 10.1136/thx.2009.124644. PMID 20335290
- [Background] Unosson J, Blomberg A, Sandstrom T, Muala A, Boman C, Nystrom R, Westerholm R, Mills NL, Newby DE, Langrish JP, Bosson JA. Exposure to wood smoke increases arterial stiffness and decreases heart rate variability in humans. Part Fibre Toxicol. 2013 Jun 6;10:20. doi: 10.1186/1743-8977-10-20. PMID 23742058
- [Background] Rudell B, Ledin MC, Hammarstrom U, Stjernberg N, Lundback B, Sandstrom T. Effects on symptoms and lung function in humans experimentally exposed to diesel exhaust. Occup Environ Med. 1996 Oct;53(10):658-62. doi: 10.1136/oem.53.10.658. PMID 8943829